CLINICAL TRIAL: NCT07168811
Title: Comparative Clinical and Radiographic Evaluation of Hyaluronic Acid, TheraCal, and Mineral Trioxide Aggregate as Pulpotomy Agents in Primary Molars: A Randomized Clinical Trial
Brief Title: Comparison of Hyaluronic Acid, TheraCal, and Mineral Trioxide Aggregate as Pulpotomy Agents in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Omaima Salah Ahmed Mohamed Elbeltagy, Doctor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1222/5298
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pulpotomies Primary Teeth; Pulp Disease, Dental
Keywords: Hyaluronic Acid; TheraCal; MTA
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Hyaluronic Acid; TheraCal; mineral trioxide aggregate

STUDY DESIGN:
Intervention Model Description: 1. Group I: Hyaluronic acid (0,5% gengigel teething). (Study group).
  2. Group II: theraCal LC. (Study group).
  3. Group III: MTA (Control group).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Operator Blinding: The operator performing the procedure will not be blinded due to the differences in handling and appearance of the materials.
  Patient and Parent Blinding: Participants and their parents/legal guardians will be blinded to the type of pulpotomy agent used. All materials will be applied under rubber dam isolation, and the clinical procedure will be standardized to avoid revealing the material identity.
  Outcome Assessor Blinding: The clinical and radiographic evaluations will be performed by a blinded, calibrated examiner who is unaware of the group assignments. The radiographs will be coded and assessed using standardized criteria to prevent bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyaluronic acid (Experimental): • After achieving complete hemostasis: Mix HA (0,5% gengigel teething) with ZO powder until a mixture, then apply it on pulp stumps.
  all teeth will be restored with glass ionomer (Prevest Denpro Micron Superior Limited, India),then a stainless steel crown (3M, ESPE, USA) to ensure proper coronal seal and long-term success, which was cemented by glass ionomer cement(Prevest Denpro Micron Luting Limited, India).
  Interventions: Procedure: Hyaluronic Acid (HA)
- TheraCal (Experimental): • After achieving complete hemostasis: TheraCal L.C will be applied directly to the radicular pulp by a disposable syringe tip and light cure will be done for 20 seconds.
  all teeth will be restored with glass ionomer (Prevest Denpro Micron Superior Limited, India),then a stainless steel crown (3M, ESPE, USA) to ensure proper coronal seal and long-term success, which was cemented by glass ionomer cement(Prevest Denpro Micron Luting Limited, India).
  Interventions: Procedure: TheraCal
- Mineral Trioxide Aggregate (Active Comparator): • After achieving complete hemostasis: mix MTA with sterile saline and put on pulp stumps. A moist cotton pellet was placed for initial setting.
  all teeth will be restored with glass ionomer (Prevest Denpro Micron Superior Limited, India),then a stainless steel crown (3M, ESPE, USA) to ensure proper coronal seal and long-term success, which was cemented by glass ionomer cement(Prevest Denpro Micron Luting Limited, India).
  Interventions: Procedure: Mineral Trioxide Aggregate

INTERVENTIONS:
Procedure: Hyaluronic Acid (HA) — • After achieving complete hemostasis:
  1. Mix HA (0,5% gengigel teething) with ZO powder until a mixture, then apply it on pulp stumps.
  2. all teeth will be restored with glass ionomer (Prevest Denpro Micron Superior Limited, India),then a stainless steel crown (3M, ESPE, USA) to ensure proper coronal seal and long-term success, which was cemented by glass ionomer cement(Prevest Denpro Micron Luting Limited, India)
  Other Names: HA Pulpotomy
  Arms: Hyaluronic acid
Procedure: TheraCal — • After achieving complete hemostasis:
  1. TheraCal L.C will be applied directly to the radicular pulp by a disposable syringe tip and light cure will be done for 20 seconds.
  2. all teeth will be restored with glass ionomer (Prevest Denpro Micron Superior Limited, India),then a stainless steel crown (3M, ESPE, USA) to ensure proper coronal seal and long-term success, which was cemented by glass ionomer cement(Prevest Denpro Micron Luting Limited, India)
  Other Names: TheraCal LC Pulpotomy
  Arms: TheraCal
Procedure: Mineral Trioxide Aggregate — • After achieving complete hemostasis:
  1. mix MTA with sterile saline and put on pulp stumps. A moist cotton pellet was placed for initial setting.
  2. all teeth will be restored with glass ionomer (Prevest Denpro Micron Superior Limited, India),then a stainless steel crown (3M, ESPE, USA) to ensure proper coronal seal and long-term success, which was cemented by glass ionomer cement(Prevest Denpro Micron Luting Limited, India)
  Other Names: MTA Pulpotomy
  Arms: Mineral Trioxide Aggregate

SUMMARY:
This randomized clinical trial aims to evaluation the clinical and radiographic outcomes of hyaluronic acid, TheraCal, and Mineral Trioxide Aggregate (MTA) when used as pulpotomy agents in primary molars.

The main question it aims to answer is:

In children with restorable mandibular second primary molars requiring pulpotomy, does the use of hyaluronic acid or TheraCal LC, compared to MTA, result in improved clinical and radiographic success rates over a 12-month follow-up period?

DETAILED DESCRIPTION:
Premature loss of primary teeth can affect occlusion development and lead to complications such as space loss and malalignment of permanent teeth. To prevent this, effective pulpotomy treatment is essential. Therefore, identifying the most suitable pulpotomy agent is crucial to retain primary teeth until their natural exfoliation.

According to MTA research, it has a high success rate as a pulpotomy agent and favors tissue regeneration while also having a good long-term prognosis, good biocompatibility, and strong sealing capacity . Among its many applications are direct pulp capping, pulpotomy, root end filling, apexification, apexogenesis, and root perforation . Low compressive strength, high pH (approximately 10.2 after setting which take 3 hours, pH increase to 12,5), high cost, short shelf life, manipulation challenges, lengthy setting time, and discoloration are some disadvantages.

TheraCal LC (Bisco, Schaumburg, IL, USA) is a novel calcium silicate-based resin-modified material designed as a liner under restorative materials to protect and stimulate the pulp in both direct and indirect pulp capping. It contains polyethylene-glycol dimethacrylate monomers, barium zirconate, and tri-calcium silicate particles. According to earlier research, the TheraCal LC material stimulated the production of secondary dentin and apatite by releasing calcium.

TheraCal provides a number of advantages over other silicate-based materials, including low solubility, easy application, good mechanical properties, setting time, adequate bonding ability, and prevention of microleakage. Commercially available as a syringe, TheraCal is user-friendly. TheraCal is a good option for kids who can't handle long visits and might eventually stop cooperating because of all these benefits.

Hyaluronic Acid (HA) is made up of polyanionic disaccharide units of N-acetyl glucosamine and glucuronic acid joined by alternating β-(1ــــ3) and β-(1ــــ4) linkages. It is a naturally occurring non-sulfated glycosaminoglycan with a high molecular weight of 4000-20,000,000 Da. It is a linear polysaccharide found in the extracellular matrix of skin, vitreous humor, embryonic mesenchyme, connective tissue, synovial fluid, and several other human tissues and organs . It is an appealing material for use in several dental operations due to its biocompatibility, regenerative qualities, and antibacterial properties .

It is used in dentistry to treat alveolar osteitis, peri-implantitis, chronic periodontitis, and gingivitis; manage wound healing following free gingival graft; control symptoms like pain, swelling, and trismus that may arise following tooth extraction; heal recurrent oral ulcers; and to manage teething symptoms. Additionally, HA is employed in research utilizing human dental pulp stem cells (hDPSCs) in an effort to offer a novel method of regenerative endodontic therapy.

So the present study will be conducted for evaluation of Hyaluronic Acid, TheraCal, and Mineral Trioxide Aggregate as Pulpotomy Agents in Primary Molars.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-8 years,
* Co-operative patient
* At least one restorable mandibular second primary molars with deep carious lesions requiring pulpotomy.
* Absence of gingival swelling or sinus tract.
* Absence of spontaneous pain.
* Absence of pain on percussion.
* Controlled bleeding.
* First treatment the tooth.
* Possibility of restoring the tooth with a stainless steel crown.
* No Radiographic evidence of changes associated with pulp degeneration, such as widening of PDL space, internal root resorption, external root resorption, inter-radicular or periapical bone destruction (radiolucency).

Exclusion Criteria:

* Swelling, sinus tract, or fistula.
* Spontaneous pain.
* Necrotic pulp, pathological mobility.
* Cases require for general anesthesia.
* A history of repeated need for analgesics.
* Patients with any systemic diseases.
* Uncontrolled bleeding.
* Selected deciduous teeth without a permanent successor

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation | 3, 6, and 12 months.
  Clinical evaluation:
  Absence of
  * Pain
  * Soft tissue swelling
  * Sinus tract
  * tenderness to percussion
  * tooth mobility
Radiographic evaluation | 3, 6, and 12 months
  Conventional radiographic evaluation:
  absence of
  * Internal resorption.
  * External resorption.
  * Periapical or furcation RL.
  * Obliteration pulp calcification.
  * Widening of periodontal space.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt

REFERENCES:
- [Background] Cameron, Angus C., and Richard P. Widmer, eds. Handbook of Pediatric Dentistry E-Book: Handbook of Pediatric Dentistry E-Book. 5th ed. Elsevier Health Sciences, 2021. P. 131.
- [Background] Khatab, Arafa, and Elsayed Mohamed Deraz. "Clinical, radiographical and histopathological evaluation of Biodentine versus formocresol in primary teeth pulpotomy." Egyptian Dental Journal 65.4-October (Orthodontics, Pediatric & Preventive Dentistry) (2019): 3199-3212
- [Background] Amrollahi N, Karimi R, Shariati F. Clinical and radiographic success of TheraCal versus Formocresol in primary teeth pulpotomy: A systematic review and meta-analysis. Saudi Dent J. 2024 Aug;36(8):1058-1065. doi: 10.1016/j.sdentj.2024.06.008. Epub 2024 Jun 6. PMID 39176161
- [Background] Jha S, Namdev R, Singhal R, Goel N, Singhal P, Rani R. Comparative Evaluation of Effectiveness of TheraCal LC, MTA, and Calcium Hydroxide in Direct Pulp Capping in Primary Molars: Randomized Clinical Study. Int J Clin Pediatr Dent. 2023 Sep;16(Suppl 2):213-219. doi: 10.5005/jp-journals-10005-2642. PMID 38078039
- [Background] Ildes GC, Sezgin BI, Vieira AR, Mentes A. A randomized clinical trial of hyaluronic acid gel pulpotomy in primary molars with 1 year follow-up. Acta Odontol Scand. 2022 May;80(4):273-280. doi: 10.1080/00016357.2021.1998612. Epub 2021 Nov 9. PMID 34752723
- [Background] Shaimaa mohamed Mahfouz; asmaa abdallah; shaimaa shaban el-desouky. "Clinical and Radiographic Evaluation of Hyaluronic Acid as a Vital Pulpotomy Medication in Primary Molars", Egyptian Dental Journal, 67, 3, 2021, 1843-1855
- [Background] Verma, Bhawna, et al. "Comparative evaluation of success of pulpotomy in primary molars treated with Formocresol, Pulpotec and Biodentine-6 month follow up study." Int J Appl Dent Sci 5 (2019): 77-82.
- [Background] Sezgin BI, Ildes Sezgin GC, Koyuncu O, Mentes A. Hyaluronic acid as a pulpotomy material in primary molars: an up to 30 months retrospective study. BMC Oral Health. 2024 Jun 12;24(1):683. doi: 10.1186/s12903-024-04405-4. PMID 38867194
- [Background] Miglani A, Vishnani R, Reche A, Buldeo J, Wadher B. Hyaluronic Acid: Exploring Its Versatile Applications in Dentistry. Cureus. 2023 Oct 2;15(10):e46349. doi: 10.7759/cureus.46349. eCollection 2023 Oct. PMID 37920632
- [Background] Casale M, Moffa A, Vella P, Sabatino L, Capuano F, Salvinelli B, Lopez MA, Carinci F, Salvinelli F. Hyaluronic acid: Perspectives in dentistry. A systematic review. Int J Immunopathol Pharmacol. 2016 Dec;29(4):572-582. doi: 10.1177/0394632016652906. Epub 2016 Jun 8. PMID 27280412
- [Background] Karadas M, Cantekin K, Gumus H, Ates SM, Duymus ZY. Evaluation of the bond strength of different adhesive agents to a resin-modified calcium silicate material (TheraCal LC). Scanning. 2016 Sep;38(5):403-411. doi: 10.1002/sca.21284. Epub 2015 Nov 10. PMID 26553783
- [Background] Tao W, Tian G, Song Q, Lv Z. Application of mineral trioxide aggregate pulpotomy in the treatment of early pulpitis of primary molars. Am J Transl Res. 2024 Jan 15;16(1):285-294. doi: 10.62347/XVVC1010. eCollection 2024. PMID 38322556
- [Background] Hamdi, Mona Nagy. "Clinical and radiographic evaluation of MTA based zinc oxide eugenol versus Formocresol pulpotomy in primary molars." Egyptian Dental Journal 69.3 (2023): 1767-1773.
- [Background] Sharaan, Marwa El-Sayed, and Mohamed Ibrahim Rabie. "Mineral Trioxide Aggregate VS Calcium Enriched Mixture molar pulpotomy: A systematic review and meta-analysis." Egyptian Dental Journal 64.1-January (Fixed Prosthodontics, Dental Materials, Conservative Dentistry & Endodontics) (2018): 363-371.